CLINICAL TRIAL: NCT01008488
Title: Is Antibiotic Therapy Mandatory for Treatment of Uncomplicated Acute Colonic Diverticulitis: a Randomized Clinical Trial
Brief Title: Antibiotic Therapy of Acute Uncomplicated Colonic Diverticulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Landstinget i Värmland (Other)
Responsible Party: Principal Investigator, achabok, MD, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVOD-D33
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Colonic Diverticulitis
Keywords: colonic diverticulitis; diverticular disease; antibiotic therapy
MeSH Terms: conditions — Diverticulitis, Colonic; Diverticular Diseases | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotic (Active Comparator)
  Interventions: Drug: Antibiotic
- No antibiotic (No Intervention)

INTERVENTIONS:
Drug: Antibiotic — Antibiotic according to local treatment routine against bowel pathogenesis
  Arms: Antibiotic

SUMMARY:
The purpose of this study is to evaluate if antibiotic therapy is necessary for treatment of uncomplicated colonic diverticulitis.

The hypothesis is that Patients with acute uncomplicated colonic diverticulitis will recover the condition without antibiotic therapy and the lack of antibiotic therapy will not lead to complications.

The patients will be randomized to conservative treatment with and without antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* adults with CT sign of acute colonic uncomplicated diverticulitis
* elevated CRP and LPK
* Temp.38c or more

Exclusion Criteria:

* patients with peritonitis, sepsis or CT- sign of complicated diverticulitis with abscesses or free abdominal air
* pregnancy
* immunological incompetence and immunosuppressive therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2002-11; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
discharge without complications +/- antibiotic therapy | Within 30 days after discharge

SECONDARY OUTCOMES:
to evaluate length of hospital stay, cost and late complications | one year after admission

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Smedh, Principal Investigator — Center of Clinical Research, Västerås
Locations (1):
- The Central Hospital, Västerås, Västmanland County, Sweden

REFERENCES:
- [Derived] Chabok A, Pahlman L, Hjern F, Haapaniemi S, Smedh K; AVOD Study Group. Randomized clinical trial of antibiotics in acute uncomplicated diverticulitis. Br J Surg. 2012 Apr;99(4):532-9. doi: 10.1002/bjs.8688. Epub 2012 Jan 30. PMID 22290281